CLINICAL TRIAL: NCT05561257
Title: A Double-blind, Placebo-controlled, 4-arm Pilot Study on the Use of Vitamin C as Add on Therapy in Patients With Acute Herpes Zoster
Brief Title: Vitamin C as add-on Therapy in Patients With Acute Herpes Zoster
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the necessary recruitment was no longer ensured and fundamental changes in the medical care of herpes zoster, which prevented the original research objectives and the feasibility of the study in the planned scope from being achieved
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 218S18VC
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (control group) (Placebo Comparator): 300 ml NaCl infusion
  Interventions: Drug: Vitamin C
- Group 2 (750 mg Vitamin C) (Experimental): 295 ml NaCl + 5 ml (750 mg) Vitamin C
  Interventions: Drug: Vitamin C
- Group 3 (7.5 g Vitamin C) (Experimental): 250 ml NaCl + 1 x 50 ml (7.5 g) Vitamin C
  Interventions: Drug: Vitamin C
- Group 4 (15 g Vitamin C) (Experimental): 200 ml NaCl + 2 x 50 ml (2 x 7.5 g) Vitamin C
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — Vitamin C

SUMMARY:
To compare the efficacy and tolerability of three different doses of Pascorbin® besides standard medication with placebo and the reduction of herpes zoster-associated clinical symptoms as an add-on therapy for patients suffering from acute herpes zoster in primary care

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients older than 18 years
2. Diagnosis of acute herpes zoster
3. Presence of at least one efflorescence
4. Peak NRS pain score ≥ 5 within the last 24h
5. Based on the appraisal of the investigator: adequate educational as well as intelligence level and communicative capacity in order to comply with the requirements of the trial
6. Written informed consent of the patient
7. Negative urine pregnancy test at the baseline visit (prior to the first infusion of study medication) for female patients of childbearing potential.
8. Women of child-bearing potential must apply during the entire duration of the trial a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1 % per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method (oestrogen and progestogen), or some intrauterine devices (IUDs) or sexual abstinence (true abstinence, only if in line with the preferred and usual lifestyle) or vasectomy of partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or post-menopausal with at least 1 year without spontaneous menses.
9. Patients are suitable for study participation according to their general medical situation

Exclusion Criteria:

1. History of oxalate-urolithiasis or nephrolithiasis
2. Current active zoster episode for more than 10 days
3. Known severe renal function impairment consistent with Kidney Disease Improving Global Outcome (KDIGO) Glomerular Filtration Rate (GFR) stages G4 and 5 (< 30 ml/min/1.73m2)
4. Known iron storage disease (e.g., thalassemia, hemochromatosis, sideroblastic anemia)
5. Known erythrocytic glucose-6-phosphate dehydrogenase deficiency (at least class 3 = 10-60% rest activity = moderate deficiency)
6. Prior vaccination with Zostavax®
7. Signs or symptoms or diagnosed complications of herpes zoster such as zoster disseminatus, zoster generalisatus, zoster meningitis, zoster encephalitis, zoster myelitis, zoster pneumonitis, acute retinal necrosis (ARN)
8. Contraindication to aciclovir treatment according to the current Summary of Product Characteristics (SmPC).
9. Any disease that may interfere with the assessment of the course of the acute varicella zoster virus reactivation e.g.

   1. dermatological diseases such as psoriasis/eczema in the area of affected dermatomes
   2. painful local or systemic diseases such as wound infection or inflammation
10. Immunodeficiency diseases, including but not limited to Human Immunodeficiency Virus (HIV)
11. Known active malignancies other than non-melanoma skin cancer (NMSC)
12. Severe uncontrolled diabetes mellitus, implanted insulin pump and severe respiratory obstructive diseases
13. Other severe concomitant diseases with severe impairment of the patient's general condition
14. History of additional herpes zoster in the last 3 months prior to baseline
15. Any of the following medication, that might interact with the study medication or interfere with its effect

    1. Intravenous virostatics like aciclovir or brivudin within 4 weeks prior to baseline
    2. Oral virostatics like aciclovir or brivudin longer than 48 hours
    3. Any supplementary ascorbic acid (vitamin C) within 4 weeks prior to baseline
    4. Long-term analgesics (including local and transdermal) for non-Herpes pain (e.g. headache, rheumatism)
    5. Intake of any analgesics longer than 3 days for treatment of the current zoster symptoms
    6. Anticonvulsive drugs (gabapentin, pregabaline) within 4 weeks prior to baseline
    7. Antiepileptic drugs (carbamazepine) within 4 weeks prior to baseline
    8. Antidepressant drugs such as tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors (SSRI/SNRI) within 4 weeks prior to baseline
    9. Neuroleptics within 2 days prior to baseline
    10. Use of topical analgesics e.g., lidocaine or capsaicin patches on the site of the current herpes zoster efflorescence within 2 days prior to baseline
16. Current therapy with immunosuppressive drugs, including but not limited to:

    1. Any systemic chemotherapeutics/cytostatic drugs
    2. Corticosteroids (> 5 mg/d prednisolone or equivalent)
    3. Methotrexate, ciclosporin, azathioprine
17. Other drugs and interventions that may cause interactions with Vitamin C, including

    1. Fluphenazine
    2. Cumarine derivates
    3. Radiation therapy
18. Nephrotoxic drugs, that may, according to the investigator's discretion, impair renal function
19. Any other non-drug treatment of the acute herpes zoster
20. Known hypersensitivity to the pharmacologic active constituents or any other ingredient of the study medication
21. Participation in another clinical trial within the last 30 days prior to inclusion, simultaneous participation in another clinical trial or previous participation in this trial.
22. Mental or physical disability or imprisonment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Mean neuropathic pain | from Baseline to V5 (day 11-13 after baseline)
  Area under the curve (AUC) of mean neuropathic pain measured by numeric rating scale (NRS) from baseline to V5

SECONDARY OUTCOMES:
Number of standard doses of permitted concomitant analgesic medication | from Baseline to V5 (day 11-13 after baseline)
  Number of standard doses of permitted concomitant analgesic medication (step 1 of analgesic potency according to WHO) from baseline to V5
  Step 1 (non-opioids: Paracetamol 500 mg, Ibuprofen 400 mg)
AUC of equianalgesic doses of permitted concomitant analgesic medication | from Baseline to V5 (day 11-13 after baseline)
  Area under the curve of equianalgesic doses of permitted concomitant analgesic medication (step 2 of analgesic potency according to WHO) from baseline to V5
  Step 2 (weak opioids: Metamizole 500 mg, Tramadol 50 mg, Tilidine/Naloxone 50 mg/4 mg)
Presence of a Post-herpetic neuralgia | at V7 (day 90 (+/- 2 days))
  Proportion of patient who developed a post-herpetic neuralgia at V7

CONTACTS AND LOCATIONS:
Overall Officials: Holger Michels, Study Director — Pascoe Pharmazeutische Praeparate GmbH; Andraes Pinter, Dr., Principal Investigator — Universitätsklinik Frankfurt am Main
Locations (3):
- Germany (3):
  - dermatologisches zentrum Bonn, Bonn, Hesse
  - Universitätsklinikum Frankfurt am Main, Frankfurt am Main, Hesse
  - Hautklinik der Universitätsmedizin Mainz KöR, Mainz, Hesse